CLINICAL TRIAL: NCT07346417
Title: Erector Spinae Plane Block Versus Quadratus Lumborum Block for Post Operative Analgesia in Pediatric Kidney Surgery
Brief Title: Erector Spinae Plane Block Versus Quadratus Lumborum Block
Acronym: ESP-QLB-Peds
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amr omar abdulrazzaq omar, Principal Investigator, Department of Anesthesia and Intensive Care, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pediatric-Block-Study-2025
Record Dates: First submitted 2025-12-25; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Kidney Diseases
Keywords: Pediatric- kidney-surgery
MeSH Terms: conditions — Kidney Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Erector spinae plane block (Experimental): Ultrasound-guided erector spinae plane block performed at the thoracic level using a multi-shot technique after completion of surgery and before extubation for pediatric kidney surgery to provide postoperative analgesia.
  Interventions: Procedure: Quadratus lumborum block teqnique; Procedure: Erector spinae plane block Technique
- Quadratus lumborum block (Active Comparator): Ultrasound-guided quadratus lumborum block performed using a multi-shot technique, after completion of surgery and before extubation of anesthesia for pediatric kidney surgery to provide postoperative analgesia.
  Interventions: Procedure: Quadratus lumborum block teqnique; Procedure: Erector spinae plane block Technique

INTERVENTIONS:
Procedure: Quadratus lumborum block teqnique — All blocks were performed under ultrasound guidance. A high-frequency linear probe was positioned in the mid-axillary line cranial to the iliac crest to identify the abdominal wall muscles (external oblique, internal oblique, and transversus abdominis). The probe was then moved dorsally until the transversus abdominis muscle became aponeurotic, which was followed medially to visualize the quadratus lumborum (QL) muscle at its attachment to the L4 transverse process adjacent to the psoas muscle.
  Using an in-plane anterior-to-posterior approach, the block needle was advanced toward the anterior border of the QL muscle. After confirming the needle tip position with a 1 ml saline test injection, 0.5 ml/kg of 0.25% bupivacaine was administered. Bilateral injections were performed for midline incisions, while unilateral injections were used for paramedian incisions.
Procedure: Erector spinae plane block Technique — Ultrasound-guided erector spinae plane block performed at the thoracic level using a single-shot technique in pediatric patients undergoing kidney surgery to provide postoperative analgesia. Local anesthetic is injected deep to the erector spinae muscle over the transverse process with expected craniocaudal spread.

SUMMARY:
To compare the efficacy and safety of ultrasound-guided ESPB versus QLB for post-operative analgesia in children undergoing kidney surgery.

DETAILED DESCRIPTION:
The management of postoperative pain in pediatric kidney surgery is a critical component of enhanced recovery and improved patient outcomes. Effective analgesia minimizes opioid consumption and their associated side effects, facilitating early mobilization and discharge. Regional anesthesia techniques have gained prominence as opioid-sparing modalities in pediatric patients, with the erector spinae plane block (ESPB) and quadratus lumborum block (QLB) increasingly used in abdominal and renal surgeries.

The erector spinae plane block is a fascial plane block targeting the dorsal rami of spinal nerves, providing extensive analgesia for thoracic and abdominal procedures. It is considered relatively easy and safe to perform under ultrasound guidance and has been associated with effective postoperative analgesia and reduced opioid requirements in pediatric renal surgery. Additional advantages include shorter block performance time and a lower incidence of postoperative nausea and vomiting compared with other regional techniques.

The quadratus lumborum block involves local anesthetic deposition near the quadratus lumborum muscle and can be performed using different approaches, such as anterior and transmuscular techniques. These approaches provide both somatic and visceral analgesia for lower abdominal and renal surgeries. Continuous quadratus lumborum block has demonstrated effective postoperative pain control, reduced need for rescue analgesia, and minimal adverse events in pediatric renal procedures. It is also recognized for its favorable safety profile and its contribution to improved quality of recovery.

Although both ESPB and QLB are effective regional techniques for pediatric postoperative analgesia, studies comparing their efficacy have reported variable results. Some investigations have shown comparable pain scores and opioid consumption between the two blocks, while others suggest potential advantages of one technique over the other in terms of analgesic duration, side-effect profile, or patient satisfaction.

Pain assessment in pediatric patients remains challenging because of differences in age, cognitive development, and communication abilities. This necessitates the use of objective pain scoring systems and careful perioperative analgesic planning. Consequently, evaluating and comparing the analgesic efficacy and safety of these two regional blocks in pediatric kidney surgery is of particular clinical importance.

The rationale of this study is to provide direct comparative evidence on the effectiveness and safety of ultrasound-guided ESPB versus QLB for postoperative analgesia in pediatric kidney surgery. Clarifying which technique offers superior analgesic control with fewer side effects may help optimize perioperative pain management protocols and improve postoperative outcomes. This study aims to assess postoperative pain scores, opioid consumption, block-related complications, and recovery quality in order to guide anesthetic decision-making in pediatric renal surgery

ELIGIBILITY:
Inclusion Criteria:

Children of both sexes, aged 2-12 years, with ASA physical status I-II scheduled for elective unilateral kidney surgery will be eligible.

Exclusion Criteria:

* Infection at the site of needle insertion
* Allergy to local anesthetics
* Parental refusal of consent

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2025-12-25 (Estimated); Primary Completion 2028-02-28 (Estimated); Study Completion 2028-03-30 (Estimated)

PRIMARY OUTCOMES:
Time to first rescue analgesia | 24 hours
  measured from extubation until the first request/administration of analgesia, in hours

SECONDARY OUTCOMES:
Total analgesic consumption | 24 hours
  Total 24-hour postoperative analgesic consumption (mg/kg paracetamol, µg/kg fentanyl).
Postoperative pain score | 24 hours
  FLACC pain score assessed at 0, 1, 2, 6, 12, and 24 hours postoperatively.
Incidence of postoperative nausea and vomiting | 24 hours
  Incidence of PONV within 24 hours postoperatively.
Block-related complications | 24 hours
  Incidence of block-related complications.
Postoperative hemodynamic stability | 24 hours
  Changes in heart rate and blood pressure >20% from baseline.
Parent satisfaction | 24 hours
  Parent satisfaction measured using a 5-point Likert scale.

REFERENCES:
- [Result] Wu X, He H, Zhao L, Zeng Z, Yuan J. Case Report: Gastric cancer with chondromyxoid matrix similar matrix-producing metaplastic breast carcinoma: report of an undescribed entity. Front Oncol. 2023 May 19;13:1087241. doi: 10.3389/fonc.2023.1087241. eCollection 2023. PMID 37274268
- [Result] Sac G, Ozulug M, Geiger MF, Freyhof J. Pseudophoxinus cilicicus, a new spring minnow from southern Anatolia (Teleostei: Leuciscidae). Zootaxa. 2019 Sep 16;4671(1):zootaxa.4671.1.8. doi: 10.11646/zootaxa.4671.1.8. PMID 31716597
- [Result] Aksu C, Gurkan Y. Ultrasound guided erector spinae block for postoperative analgesia in pediatric nephrectomy surgeries. J Clin Anesth. 2018 Mar;45:35-36. doi: 10.1016/j.jclinane.2017.12.021. Epub 2017 Dec 20. No abstract available. PMID 29274546
- [Result] Wu L, Zhang W, Wei Y, Zhang D. Comparison of the analgesic effects of ultrasound-guided erector spinae plane block and quadratus lumborum block: a systematic review and meta-analysis. Front Pharmacol. 2025 Aug 1;16:1640135. doi: 10.3389/fphar.2025.1640135. eCollection 2025. PMID 40822461
- [Result] Aksoy M, Aksoy AN, Yilmaz EPT, Senocak GNC, Dostbil A, Ozkan H. The effectiveness of erector spina plane, quadratus lumborum blocks, and intrathecal morphine for analgesia after cesarean: a randomized study. Rev Assoc Med Bras (1992). 2023 Nov 13;69(12):e20230867. doi: 10.1590/1806-9282.20230867. eCollection 2023. PMID 37971133
- [Result] Zhang M, Zhao S, Song S, Zhou H, Li M, Su P, Xu G. Comparative analgesic efficacy of erector spinae plane block versus quadratus lumborum block in laparoscopic renal cancer surgery: a double-blind randomized trial. Transl Androl Urol. 2025 Jul 30;14(7):2029-2042. doi: 10.21037/tau-2025-71. Epub 2025 Jul 28. PMID 40800097
- [Result] An Y, Li L, Li Z, Lan F, Wang T, Ou T, Liang C, Wang P, Jia X, Song H, Cui K, Luo H, Zhao L. Anterior quadratus lumborum block is superior to erector spinae plane block for analgesia after renal transplantation: a randomized controlled trial. BMC Anesthesiol. 2025 Jul 10;25(1):343. doi: 10.1186/s12871-025-03209-5. PMID 40640721
- [Result] Wu H, Huang J. Quadratus lumborum block versus caudal block in paediatric surgeries: a protocol for systematic review and meta-analysis. BMJ Open. 2025 May 28;15(5):e100085. doi: 10.1136/bmjopen-2025-100085. PMID 40441771
- [Result] Kayumova PM, Giyasov SI, Krasnenkova MB, Musabaev AN. Erector Spinae Plane block: evaluation of its efficacy as a component of multimodal anaesthesia in open kidney surgery. Urology Herald. 2024;12(1):36-44.
- [Result] Kambey BI, Ramlan AAW, Rahendra R, Selene NB. Ultrasonogram-Guided Continuous Quadratus Lumborum Block as Pain Management in Pediatric Kidney Transplant Recipients: A Case Series. Exp Clin Transplant. 2025 Jan;23(1):72-77. doi: 10.6002/ect.2024.0205. PMID 39918196
- [Result] Capuano P, Burgio G, Abbate S, Ranucci G, Bici K, Cintorino D, Arcadipane A, Martucci G. Continuous Erector Spinae Plane Block for Pain Management in a Pediatric Kidney Transplant Recipient: A Case Report and Review of the Current Literature. J Clin Med. 2024 Feb 17;13(4):1128. doi: 10.3390/jcm13041128. PMID 38398441